CLINICAL TRIAL: NCT03414099
Title: Ketum and Pain Tolerence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Vicknasingam B Kasinather, Professor, Universiti Sains Malaysia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: USM/JEPeM/17050243
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Pain
Keywords: Pain; Kratom; Ketum; mitragynine
MeSH Terms: conditions — Pain | interventions — mitragynine

STUDY DESIGN:
Intervention Model Description: Within-subject, repeated measures
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Ketum and placebo drinks will be matched for taste and appearence. Each study participant will receive a sequence of ketum and placebo drinks in random order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketum (Experimental): Each participant will consume a sequence of active ketum or placebo drinks. Pain tolerance will be measured using the cold pressor task after consuming each drink.
  Interventions: Drug: Ketum
- Placebo (Placebo Comparator): Each participant will consume a sequence of active ketum or placebo drinks. Pain tolerance will be measured using the cold pressor task after consuming each drink.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketum — Ketum (Mitragyna speciosa) is an indigenous plant of Southeast Asia reported to have medicinal value in traditional culture
  Other Names: Kratom
  Arms: Ketum
Drug: Placebo — Placebo drink matched for taste and appereance
  Arms: Placebo

SUMMARY:
The study aim is to evaluate potential analgesic properties of ketum using the cold pressor task.

DETAILED DESCRIPTION:
Participants in the proposed study will be individuals who report consuming ketum more than once a day, daily for the past 12 months. The study is a placebo-controlled, double-blind within-subject repeated mesaures design. Participants will ingest a sequence of ketum and placebo drinks prepared by pharmacologists at USM Centre for Drug Research and their pain tolerance will be measured by the cold pressor task after ingesting ketum or placebo.

ELIGIBILITY:
Inclusion Criteria: Individuals who report drinking ketum decoction more than once a day, daily for the past 12 months.

-

Exclusion Criteria: (1) tested positive for illicit drug use including morphine, cannabis, methamphetamine, amphetamine, methadone, benzodiazepine and ketamine; (2) have current or previous history of psychological or neurological problems (self-report); (3) have current or previous alcohol use history (self-report); (4) HIV infections; (5) history of chronic liver disease (e.g. cirrhosis, hepatitis A, B, C, etc.) 6) non-alcoholic fatty liver disease; (7) history of coronary heart disease and diabetes; (8) existing chronic pain condition and (9) history of psychiatric disorders. Exclusion criteria for female particiapns: (1) pregnancy, (2) nursing.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain tolerance | 3 hours
  The duration (seconds) participants can keep their hands immersed in the water bath

CONTACTS AND LOCATIONS:
Overall Officials: Vicknasingam Kasinather, PhD, Principal Investigator — Director
Locations (1):
- Centre for Drug Research, Univerisiti Sains Malaysia, George Town, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No